CLINICAL TRIAL: NCT01483105
Title: DVD-Based Training Program in Self-Hypnosis for Children: A Randomized Clinical Trial
Brief Title: DVD-Based Training Program in Self-Hypnosis for Children
Acronym: VCUG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, David Spiegel, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6970
Record Dates: First submitted 2011-11-18; First posted 2011-12-01 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Vesicoureteral Reflux
Keywords: VCUG; Child; Hypnosis; Relaxation; Voiding cystourethrography
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DVD self-hypnosis (Experimental): This group will receive standard care, and parents/children in this group will receive in the mail a set of questionnaires and the DVD self-hypnosis training program. Parents will be asked to review these materials and practice the training at home with their children for one week leading up to the procedure Parents will also be asked to try to use these techniques with their child during his or her upcoming VCUG procedure.
  Interventions: Behavioral: DVD Self-Hypnosis Training Program
- Standard care (No Intervention): Children in this arm will receive standard care and parents/children will be mailed a set of questionnaires to complete before and after your child's upcoming VCUG.

INTERVENTIONS:
Behavioral: DVD Self-Hypnosis Training Program — The DVD training program contains instructional materials developed by an experienced psychiatrist and psychologist at the Department of Psychiatry at Stanford University School of Medicine. Parents will be instructed to review these materials, watch the DVD, and practice the self-hypnosis exercises every day for a week with their child prior to the upcoming procedure. Parents are encouraged to practice self-hypnosis during their child's VCUG procedure.
  Arms: DVD self-hypnosis

SUMMARY:
The proposed study is designed to utilize a self-hypnosis DVD home-training program for parents to use with their children to teach self-hypnosis techniques for inducing relaxation and hypnotic analgesia. These relaxation techniques can be employed to manage anticipatory anxiety, distress, and pain during an invasive medical procedure, for example, voiding cystourethrography (VCUG). The study will examine the efficacy of this intervention for children undergoing VCUG procedures.

DETAILED DESCRIPTION:
Pediatric care professionals and parents seek safe ways to make invasive medical procedures less stressful and traumatic for children. However, for unpleasant procedures that require child cooperation, this task becomes difficult. Home-training in self-hypnotic relaxation may provide an inexpensive, yet systematic method for improving the overall medical care of children undergoing invasive medical procedures. The proposed study is designed to utilize a self-hypnosis DVD home-training program for parents to use with their children to teach self-hypnosis techniques for inducing relaxation and hypnotic analgesia. The study will examine the efficacy of this intervention for children undergoing urethral catheterization for VCUG procedures. Parents will be instructed to watch the DVD and practice the self-hypnosis exercises every day for a week with their child prior to the upcoming procedure. Parents are encouraged to practice self-hypnosis during their child's VCUG procedure. Both parents and children will be asked to complete a series of questionnaires before and following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Child and participating parent have assented (child) or consented (parent) to participate
* Both child and parent are English-speaking
* Child has undergone at least one previous VCUG
* Child was at least 4 years of age at the time of the most recent VCUG
* Parent reports child experienced some difficulty (e.g., at least some crying, pain, or fear) during that earlier procedure.

Exclusion Criteria:

* Child and participating parent have not assented (child) or consented (parent) to participate
* Either child or parent are not English-speaking
* Child has not undergone at least one previous VCUG
* Child was under 4 years of age at the time of the most recent VCUG
* Parent reports child did not experience difficulty (e.g., at least some crying, pain, or fear) during that earlier procedure.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07-06 (Actual); Study Completion 2012-07-06 (Actual)

PRIMARY OUTCOMES:
Distress: Child Self-Report | Same day - one week after procedure
  Crying will be assessed by having the child point to a picture on a continuous visual analog scale of 6 different faces representing increasing levels of distress, ranging from a smiling face to a face crying intensely.
Distress: Parent Report | Same day - one week after procedure
  Parent assessments of child distress (fear, pain, and crying)and overall trauma will be completed on 5-point scales, ranging from "not at all" to "extremely". Parents will also rate of how traumatic the present VCUG procedure was compared with the previous one was completed on a 6-point scale ranging from "much less traumatic" to "much more traumatic."
Distress: Observational Ratings | Same day - while the child is undergoing the VCUG procedure. Time can range from minutes - hours of observation.
  A research associate will rate the child's distress from the time he or she enters the procedure room until the procedure is completed. A modified 8-point version of the Torrance Global Mood Scale will be used.

SECONDARY OUTCOMES:
Difficulty of Procedure: Medical Staff Ratings | Directly following procedure - up to 30 minutes following the end of procedure.
  Immediately after the procedure, the attending radiologist and the technician each will be asked to rate the degree of difficulty of conducting the procedure. Staff will be asked to make the ratings with respect to children of similar ages on a 7-point scale ranging from "far easier" to "far more difficult."
Anxiety: Parent Self-Report | Directly following procedure - up to 30 minutes following the end of procedure.
  Parents will complete the State-Trait Anxiety Inventory (Spielberger, 1970) immediately following the procedure.
Parent Confidence | Directly following procedure - 1 week
  Parent confidence in helping their child through the VCUG procedure will be assessed immediately following the procedure up to 1 week.
DVD Evaluation | Same day - 3 months following procedure
  The DVD Evaluation form will ask parents to evaluate the DVD-based training program.
Duration of Procedure | Same day - Time can range from minutes - hours of observation.
  Time in minutes of the VCUG procedure will be recorded from when the child first enters the room to when the child is told the procedure is over.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University School of Medicine, Department of Psychiatry and Behavioral Sciences; Linda M. Shortliffe, M.D., Study Director — Stanford University School of Medicine, Pediatric Urology
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] Butler LD, Symons BK, Henderson SL, Shortliffe LD, Spiegel D. Hypnosis reduces distress and duration of an invasive medical procedure for children. Pediatrics. 2005 Jan;115(1):e77-85. doi: 10.1542/peds.2004-0818. PMID 15629969
- See also: DVD study screen — https://stanfordmedicine.qualtrics.com/SE/?SID=SV_e9Rm0i6H0uyxiw4